CLINICAL TRIAL: NCT06888557
Title: A Proactive Patient-centered Interactive Smartphone-based Self-Management Support Program for Patients With Chronic Obstructive Pulmonary Disease - A Pragmatic Randomized Controlled Trial With Mixed-method Evaluation
Brief Title: Smartphone-based Self-Management Support Program to Enhance Quality of Life in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: United Christian Hospital (Other); Queen Mary Hospital, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Agnes LAI Yuen Kwan, Associate Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE-SF2023/04
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; self-management; digital; mobile; smartphone; QOL; quality of life; mixed-method
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The General Hygiene (GHI) group (No Intervention): The General Hygiene (GHI) group will not receive any intervention within the study period other than some general hygiene information, and will not join the mutual support group.
- The Intervention (3S-C) group (Active Comparator): The 3S-C intervention group will receive a smartphone-based self-management support program for them to motivate, actively engage and empower self-management, supplement current service, and provide remote continuous support within the study period.
  Interventions: Behavioral: Smartphone-based self-management support program ( 3S-C)

INTERVENTIONS:
Behavioral: Smartphone-based self-management support program ( 3S-C) — The 3S-C include: (1) two 30-minute individual sessions ; (2) a set of instant messages, 10-minute telephone-delivered health coaching ; (3) continuous personalized chat-based messaging, phone call support, and hotline service ; (4) an e-platform for goal setting and self-monitoring ; (5) A mutual support group session.
  Arms: The Intervention (3S-C) group

SUMMARY:
The goal of this study is to find out if a smartphone-based program (called 3S-C) can help people with COPD live better, healthier lives. It will also look at how the program affects their knowledge, habits, and overall health.

The main questions the study wants to answer are:

* Does the 3S-C program help people with COPD feel better and improve their quality of life?
* Does it help them understand and manage their condition better?
* Does it improve their health, such as reducing breathing problems or making it easier to sleep?
* Can it reduce the need for hospital visits or other healthcare?

Participants will be split into two groups:

The 3S-C group: They will use the smartphone-based program, which includes: (i) Two short individual sessions to motivate them, (ii) helpful messages sent through apps like WhatsApp or WeChat; (iii) support through personalized messaging, phone calls, and a hotline; (iv) an online platform to track their health; and (v) a group session to connect with other COPD patients.

The general hygiene (control) group: They will get information about staying healthy, such as tips on hand washing, food safety, keeping their home clean, and better sleep habits.

What will participants do?

Take part in the study for 12 months. visit the clinic for checkups and complete surveys and simple fitness tests at the start, after 4 months, and after 12 months.

Researchers will check if the 3S-C program improves:

* quality of life and how well people manage their condition.
* habits like taking medication on time, exercising, eating well, or quitting smoking.
* health outcomes like breathing, sleep, or feeling less anxious or depressed.

This study will compare the 3S-C program to general hygiene tips to see if using a smartphone can make living with COPD easier and healthier.

DETAILED DESCRIPTION:
COPD is a progressive condition that worsens with age, significantly impacting patients, families, and society due to declining health status, reduced quality of life, and high healthcare utilization. Quality of life impairment remains a critical issue for individuals with COPD.

This assessor-blinded, two-armed randomized controlled trial, with a 12-month follow-up, will recruit 130 eligible patients who will be randomized in blocks of 4-6 into either the intervention group (n=65) or the control group (n=65). The intervention group will receive the 3S-C smartphone-based self-management support program, while the control group will receive general hygiene (GH) information.

The 3S-C program is designed to enhance patients' knowledge, skills, confidence, and self-management of their illness. It includes two 30-minute motivational enhancement sessions, staged WhatsApp/WeChat messages, personalized chat-based support (messaging, phone calls, and hotline services), an e-platform for self-monitoring, and a mutual support group session. In contrast, the GH program provides education on personal hygiene (e.g., hand washing), food hygiene (e.g., safe food storage), environmental hygiene (e.g., pest control), and sleep hygiene (e.g., avoiding caffeine before bedtime).

The primary objective of this trial is to evaluate the impact of the 3S-C program on quality of life in COPD patients. Secondary outcomes include improvements in health-related cognition (knowledge, self-efficacy, and acceptance of illness), behavior (medication adherence, inhalation technique, physical activity, dietary habits, and smoking cessation), clinical outcomes (dyspnea, exacerbations, exercise capacity, sleep quality, and mental health), and healthcare utilization (frequency of hospital visits and emergency care).

Data will be collected at baseline, 4 months, and 12 months through surveys and simple fitness tests. Additionally, focus group interviews will be conducted. This study will determine if the 3S-C program effectively improves quality of life and health outcomes for COPD patients while reducing healthcare utilization. If successful, the 3S-C program could provide a scalable, low-cost solution to enhance COPD management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and above
* Confirmed diagnosis of COPD
* Had COPD acute exacerbation in prior 6 months that required hospitalization, medical intervention or seek medical consultation
* Mentally, cognitively and physically fit to join as determined by the doctor in-charge and responsible clinical investigators
* Can speak and read Chinese
* Completion of the Physical Activity Readiness Questionnaire
* Has a smartphone with WhatsApp or WeChat

Exclusion Criteria:

* Have other significant lung disease or Class 4 heart failure [defined by the New York Heart Association classification]
* Serious active infection
* Inability to walk
* Unstable psychiatric illness

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Baseline, month 4
  Measured by an 8-item COPD Assessment Test (CAT). Each item score ranges from 0 to 5. The total score ranges from a minimum of 0 to a maximum of 40. Higher scores denote a more severe impact of COPD on a patient's life. The difference between stable and exacerbation patients was five units. No target score represents the best achievable outcome.

SECONDARY OUTCOMES:
Change in quality of life | Baseline, month 12
  Measured by an 8-item COPD Assessment Test (CAT). Each item score ranges from 0 to 5. The total score ranges from a minimum of 0 to a maximum of 40. Higher scores denote a more severe impact of COPD on a patient's life. The difference between stable and exacerbation patients was five units. No target score represents the best achievable outcome.
Change in patient activation | Baseline, month 4 and 12
  Measured by a 13-item Patient Activation Measure with a 5-point Likert response scale from 0 to 4. Raw scores are transformed to a scale of 0-100 with higher scores indicating a higher activation in self-management.
Change in self-efficacy for self-management | Baseline, month 4 and 12
  Measured by a 6-item Stanford self-efficacy scale ranging from 1 to 10 for each item. The score for the scale is the mean of the six items. Minimum score is 1 and the maximum score is 10. If more than two items are missing, do not score the scale. Higher number indicates higher self-efficacy.
Change in acceptance of illness | Baseline, month 4 and 12
  Measured by an 8-item Acceptance of Illness Scale. The scale consists of 8 statements expressing specific difficulties and limitations caused by the disease. Each item ranges from 1 to 5. The total score with a minimum of 8 and a maximum of 40.
Change in medication adherence | Baseline, month 4 and 12
  Medication adherence was measured by a checklist and was calculated as a ratio of the number of doses taken to the number of doses prescribed;
Change in PAP treatment adherence (optional for those using PAP machine) | Baseline, month 4 and 12
  Information on the number of days using the PAP and total duration of machine used per day in the past 3 month will be retrieved from built-in machine record.
Change in inhaler technique | Baseline, month 4 and 12
  Inhaler technique assessed by a 10-item checklist with answer of "Yes" or "No" . The proportion of correctness will be calculated the number of correct step divided by the number of step expected to perform.
Change in physical activity level | Baseline, month 4 and 12
  Measured the days and duration of physical activity level (light, moderate and vigorous) and sitting time in the past 7 days by the International Physical Activity Questionnaire (short version) with 4 questions.
Change in dietary habit | Baseline, month 4 and 12
  Measured by 10-item dietary intake and practice outcome based questions
Change in dyspnea severity | Baseline, month 4 and 12
  Measured by a 1-item MRC dyspnoea scale ranging from 1 to 10. Higher score shows more dyspnoea
Change in exacerbation | Baseline, month 4 and 12
  The number of episode of exacerbation will be reported by patients (including use of self-help packs, need medical consultations or medical treatment for his/her shortness of breath).
Change in health status | Baseline, month 4 and 12
  Measured by 5-item EuroQol-5D Questionnaire. Each item is a different dimension that ranges from level 1-5, a higher level indicates a more severe level of perceived problem of that dimension.
Change in subjective happiness | Baseline, month 4 and 12
  Measured by 4-item Subjective Happiness Scale with a 7-point Likert scale. Total scores range from 4 to 28. The highest scores reflect greater happiness.
Change in sleep quality | Baseline, month 4 and 12
  Measured by 7-item Severe Insomnia Index. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 28. The higher scores the greater severity of insomnia.
Health care resource utilization | Baseline, month 4 and 12
  assessed by number of hospitalizations, primary and secondary care visits, number of unscheduled admissions; and length of hospital stay.
Change in anxiety symptoms | Baseline, month 4 and 12
  Measured by a 7-item Generalised Anxiety Disorder Assessment. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 21. The higher scores the greater severity of anxiety symptoms
Change in functional exercise capacity | Baseline, month 4 and 12
  Measured by a 6-minute walk test. The distance of participant walked with the instructions to walk back and forth at their own pace to a designated spot for 6 minutes.
Change in grip strength | Baseline, month 4 and 12
  measured by dynamometer
Change in lower limb muscle strength | Baseline, month 4 and 12
  Measured by a 30-second chair stand test. The number of participant stood up repeatedly from a chair for 30 seconds.
Change in depression symptoms | Baseline, month 4 and 12
  Measured by a 9-item Patient Health Questionnaire. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 27. The higher scores the greater severity of depression symptoms.
Change in smoking and drinking habits | Baseline, month 4 and 12
  Measured by self-reported smoking and drinking frequency
Change in objective activity level | Baseline, month 4 and 12
  Measured by activity tracker for 7 days to record the activity and sleep patterns

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (3):
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - Queen Elizbeth Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao H, Kanda K. Translation and validation of the standard Chinese version of the EORTC QLQ-C30. Qual Life Res. 2000 Mar;9(2):129-37. doi: 10.1023/a:1008981520920. PMID 10983477
- [Background] Ansari S, Hosseinzadeh H, Dennis S, Zwar N. Activating primary care COPD patients with multi-morbidity through tailored self-management support. NPJ Prim Care Respir Med. 2020 Apr 3;30(1):12. doi: 10.1038/s41533-020-0171-5. PMID 32245961
- [Background] Kjellsdotter A, Andersson S, Berglund M. Together for the Future - Development of a Digital Website to Support Chronic Obstructive Pulmonary Disease Self-Management: A Qualitative Study. J Multidiscip Healthc. 2021 Apr 6;14:757-766. doi: 10.2147/JMDH.S302013. eCollection 2021. PMID 33854327
- [Background] Slevin P, Kessie T, Cullen J, Butler MW, Donnelly SC, Caulfield B. A qualitative study of chronic obstructive pulmonary disease patient perceptions of the barriers and facilitators to adopting digital health technology. Digit Health. 2019 Aug 25;5:2055207619871729. doi: 10.1177/2055207619871729. eCollection 2019 Jan-Dec. PMID 31489206
- [Background] Slevin P, Kessie T, Cullen J, Butler MW, Donnelly SC, Caulfield B. Exploring the potential benefits of digital health technology for the management of COPD: a qualitative study of patient perceptions. ERJ Open Res. 2019 May 10;5(2):00239-2018. doi: 10.1183/23120541.00239-2018. eCollection 2019 Apr. PMID 31111039
- [Background] Shaw G, Whelan ME, Armitage LC, Roberts N, Farmer AJ. Are COPD self-management mobile applications effective? A systematic review and meta-analysis. NPJ Prim Care Respir Med. 2020 Apr 1;30(1):11. doi: 10.1038/s41533-020-0167-1. PMID 32238810
- [Background] McCabe C, McCann M, Brady AM. Computer and mobile technology interventions for self-management in chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 May 23;5(5):CD011425. doi: 10.1002/14651858.CD011425.pub2. PMID 28535331
- [Background] Ding H, Fatehi F, Maiorana A, Bashi N, Hu W, Edwards I. Digital health for COPD care: the current state of play. J Thorac Dis. 2019 Oct;11(Suppl 17):S2210-S2220. doi: 10.21037/jtd.2019.10.17. PMID 31737348
- [Background] Rogliani P, Ora J, Puxeddu E, Matera MG, Cazzola M. Adherence to COPD treatment: Myth and reality. Respir Med. 2017 Aug;129:117-123. doi: 10.1016/j.rmed.2017.06.007. Epub 2017 Jun 13. PMID 28732818
- [Background] Miravitlles M, Ribera A. Understanding the impact of symptoms on the burden of COPD. Respir Res. 2017 Apr 21;18(1):67. doi: 10.1186/s12931-017-0548-3. PMID 28431503